CLINICAL TRIAL: NCT01892501
Title: Feasibility Study on the Contribution of Guided Puncture With Echoendoscopy in Evaluation of Hypermetabolic Lymphadenopathy Mediastinum Lower, Rear and Middle, Detected in PET-CT to 18 FDG (PET)
Brief Title: Feasibility Study on the Contribution of Guided Puncture With Echoendoscopy
Acronym: APOGEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IB 2012-01
Record Dates: First submitted 2013-06-26; First posted 2013-07-04 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2021-04

CONDITIONS: Hypermetabolic Lymphadenopathy Mediastinum Lower, Posterior and Middle, Detected by PET-CT With 18F-FDG (PET)
Keywords: Mediastinal lymphadenopathy; PET CT to 18FDG; EUS
MeSH Terms: interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hypermetabolic mediastinal lymph nodes in PET, (Other): hypermetabolic mediastinal lymph nodes in PET,in a context of New cancer or cancer recurrence.
  Interventions: Procedure: Guided punction of mediastinal lymphadenopathy by echoendoscopy; Device: PET scan

INTERVENTIONS:
Procedure: Guided punction of mediastinal lymphadenopathy by echoendoscopy — EUS (by oesophageal) is performed within a maximum period of six weeks after the PET scan, under general anesthesia and endoscopic control, with a disposable 19-gauge needle (EchoTip, Cook Endoscopy) and 3 passes of the needle ganglion.
  Pathological samples are taken :
  3 tubes collected by node (one tube per needle pass), in most cases, only one node will be taken.
Device: PET scan — The benefits of combined PET and punction EUS for the diagnosis and subsequent therapeutic management should be evaluated in these different contexts

SUMMARY:
Impact of screening nodes mediastinal by PET, at different times of the management of cancer disease, remain unclear.

Benefits of combined PET and puncture with echoendoscopy for the diagnosis subsequent therapeutic management should be evaluated in these different contexts.

We would like to demonstrate the clinical utility of this association to replace more invasive diagnostic procedures and to assess the impact of the puncture on a possible modification of the therapeutic management.

It is a single center prospective diagnostic assessment

DETAILED DESCRIPTION:
Main objective :

Assess the performance (in terms of sensitivity) of guided punction by echoendoscopy in the characterization of hypermetabolic mediastinal lymph nodes in PET, in a context of New cancer or cancer recurrence.

Conduct of the study :

When a patient has had a PET scan showing a hypermetabolic or mediastinal lymph nodes in the lower, middle or posterior, his case is presented in a multidisciplinary meeting (PCR # 1), with definition of diagnostic strategy:

Approved indication is achieve a biopsy surgically to have a histological documentation of mediastinal lymph nodes with obvious impact on treatment decisions.

We distinguish two groups of patients based on the feasibility of the surgical procedure:

1. Group A biopsy is surgically feasible
2. Group B: biopsy by surgery can not be performed (against medical contraindications or anesthetics) at that moment, definition of therapeutic strategy that was decided in the absence of histological documentation:

   * Surgery outset
   * Chemotherapy or other oncological treatment
   * Supports non-oncological if benign disease suspected
   * No treatment.

EUS is performed by oesophageal for two patient groups for the two groups of patients (within a maximum period of six weeks after the PET scan), under general anesthesia and endoscopic control.

According the pathological findings, the therapeutic strategy is defined in a second PCR (PCR # 2), to assess the impact of the puncture:

* Surgery outset
* Chemotherapy or other oncological treatment
* Supports non-oncological when benign pathology documented
* No treatment
* Selecting another surgical diagnostic procedure (non-contributory income).

A patient monitoring will be conducted for 12 months. The clinical and radiological data carried over the standard of care of the patient will be collected. Achieving a thoracoabdominopelvic scanner (TAP) at 1 year to characterize the evolution of the disease marks the end of the study for the patient.

For the patients who have had a negative biopsy, monitoring will involve a scanner TAP 6 month and 12 month then consultation with the oncologist.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients who have had PET showing one or more hypermetabolic lymphadenopathy in middle mediastinum and/or lower and/or posterior, and requiring diagnostic certainty for support.
2. PET scans performed in these particulars :

   * Pre-treatment assessment of thoracic or extra-thoracic malignancies (patients without a history of cancer).
   * Evaluation of response to treatment referred to oncological.
   * Suspicion of relapse in patients with a personal history of thoracic or extra-thoracic malignancies.
3. PET, the result is positive :

   * For above-centimeter lymph node short axis: greater result than or equal to the background hepatic noise.
   * For sub-centimeter lymph node small axis : greater result than the background hepatic noise
4. Patient with indication of diagnostic procedure surgically (whether realized or not)
5. Lymph node(s) available(s) puncture by EUS esophageal, so for a technically feasible for esophageal puncture (without vascular recusants structures)
6. Age ≥ 18 years.
7. PET scan performed within 6 weeks before EUS
8. Platelets ≥ 70 000/mm3; TP ≥ 60%.
9. Patient of childbearing age with negative pregnancy test and / or a contraception.
10. Patient gave informed consent signed.
11. Patient affiliated to a social security scheme.

Exclusion Criteria:

* Contra-indication (s) Director (s) to achieve a EUS.
* Balance adverse anesthetic (not allowing a general anesthetic).
* Esophageal stenosis.
* Coagulation disorders.
* Pregnant or lactating women.
* Unable to undergo medical monitoring test for geographical, social or psychological reasons.
* Private patient freedom and major subject of a measure of legal protection or unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Insitut Bergonie, Bordeaux, Grionde, France

REFERENCES:
- [Background] Bechade D, Bellera C, Gauquelin L, Soubeyran I, McKelvie-Sebileau P, Debled M, Chomy F, Roubaud G, Fonck M, Pernot S, Roch A, Cazeau AL. Diagnostic accuracy and clinical impact of endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) in Positron Emission Tomography - Computed Tomography (PET-CT)-positive mediastinal lymphadenopathies in patients with thoracic or extra-thoracic malignancies. Clin Res Hepatol Gastroenterol. 2022 May;46(5):101912. doi: 10.1016/j.clinre.2022.101912. Epub 2022 Mar 25. PMID 35341993

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypermetabolic Mediastinal Lymph Nodes in PET,: Hypermetabolic mediastinal lymph nodes in PET,in a context of New cancer or cancer recurrence.
  Guided punction of mediastinal lymphadenopathy by echoendoscopy: EUS (by oesophageal) is performed within a maximum period of six weeks after the PET scan, under general anesthesia and endoscopic control, with a disposable 19-gauge needle (EchoTip, Cook Endoscopy) and 3 passes of the needle ganglion.
  Pathological samples are taken :
  3 tubes collected by node (one tube per needle pass), in most cases, only one node will be taken.
  PET scan: The benefits of combined PET and punction EUS for the diagnosis and subsequent therapeutic management should be evaluated in these different contexts
Period: Overall Study
Arm/Group | Hypermetabolic Mediastinal Lymph Nodes in PET,
Started | 75
Group A : Biopsy Surgically Possible (Eligible for surgical procedure : Patients with no major protocol violation or medical contraindication) | 72
Group B : Biopsy Not Surgically Possible (No eligible for surgical procedure : major protocol deviations or medical contraindication) | 3
Completed | 47
Not Completed | 28
Not completed — Protocol Violation | 2
Not completed — Puncture not carried out | 9
Not completed — Radiological monitoring not carried out | 5
Not completed — Non-contributory histological result | 12

BASELINE CHARACTERISTICS:
Arm/Group | Hypermetabolic Mediastinal Lymph Nodes in PET,
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.01 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 166.97 (8.67)
Weight [Mean (Standard Deviation); unit: kg] | 72.53 (16.46)
Therapeutic strategy (absence of documentation) [Count of Participants; unit: Participants] — Therapeutic strategy before the results of the endoscopy
  Participants
    Not available | 1
    Surgery right from the start | 4
    Chemotherapy or other carcinological treatment | 54
    Non-carcinological management in case of documented benign pathology | 12
    No treatment | 4
Therapeutic strategy after documentation [Count of Participants; unit: Participants] — Therapeutic strategy after documentation (results of the endoscopy) for patients with available data Population: missing data
  Participants
    number analyzed (Participants) | 41
    Missing | 8
    Chemotherapy or other carcinological treatment | 20
    No treatment | 13
T status (Classification of Malignant Tumors) [Count of Participants; unit: Participants] — The letter "T" corresponds to the initial tumour. T classification is rated from TX (when primary lesion is not determined not assessable) or T0 (when the primary lesion is not localised) to T4 for the most extensive tumours. Population: missing data
  Participants
    number analyzed (Participants) | 37
    T0 | 1
    T1 | 7
    T2 | 9
    T3 | 13
    T4 | 5
    TX | 2
N status (Classification of Malignant Tumors) [Count of Participants; unit: Participants] — N means lymph nodes. It describes the spread of cancer to the lymph nodes surrounding the organ. N0 means that the cancer has not spread to any nearby lymph nodes. N1, N2 or N3 means that the cancer has spread to the lymph nodes. N+ means presence of lymph node. NX means non-assessable adenopathies. Population: Patients with available TNM status
  Participants
    number analyzed (Participants) | 37
    Missing | 6
    N0 | 11
    N+ | 17
    NX | 3
M status (Classification of Malignant Tumors) [Count of Participants; unit: Participants] — M classification is rated M0 in the absence of known metastases, M1 in their presence, MX when metastases are not assessable. Population: Patients with available TNM status
  Participants
    number analyzed (Participants) | 37
    Missing | 5
    M0 | 17
    M1 | 2
    Could not be evaluated for distant metastases | 13
Total number of lymph nodes per patient [Median (Full Range); unit: lymph nodes] | 3.00 [1.00 to 5.00]

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Endoscopic Ultrasound-guided (EUS-guided) Puncture
Description: The performance of EUS-guided biopsy has been evaluated in terms of sensitivity. EUS-guided was performed after detection of lymph nodes with positron emission tomography (PET). In most cases, only one lymph node is taken and performance analysis will be done by patient and not by injury.
  PET, the reference technique (gold standard), is followed for 12 months. Sensitivity is the rate of subjects with a diagnosis of malignancy (excluding the results atypical / suspicious or non-contributory) according the results of EUS among all subjects with a neoplastic disease by the gold reference.
  To sum up , the sensitivity corresponds to the rate of patients detected as "malignant" with the new technique (EUS-guided), among the patients detected as "malignant" at the reference PET examination (12 months assessment).
Time Frame: 12 months
Population: Patient eligible and evaluable for primary endpoint (N=47) (excluded patients with non-contributory histological results, puncture not carried out, radiological monitoring not carried out)
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Hypermetabolic Mediastinal Lymph Nodes in PET,
Number analyzed (Participants) | 47
percentage | 93 [76 to 99]

2. Secondary Outcome: Negative Predictive Value
Description: The negative predictive value of EUS-guided biopsy has been evaluated by the rate of subjects with a diagnosis of benign pathology according the gold standard (PET) among all subjects for wich EUS reveal a benign pathology (excluding atypical/suspects findings or non contributory)
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Hypermetabolic Mediastinal Lymph Nodes in PET,
Number analyzed (Participants) | 47
percentage | 90 [71 to 99]

3. Secondary Outcome: Matching Between Therapeutic Strategies RCP1/RCP2
Description: Impact of the management of patient :
  Concordance between therapeutic strategies before the results of the endoscopy (Multidisciplinary consultation meeting 1 (RCP1) in absence of documentation) and after the results of endoscopy (Multidisciplinary consultation meeting 2 (RCP2) post-documentation) for the eligible and evaluable population
Time Frame: 12 months
Population: Patients eligible and evaluable with available pre (before endoscopy results) AND post documentation (after endoscopy results) therapeutic strategies.
  Of note, 6 patients without therapeutic strategies after endoscopy results.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Hypermetabolic Mediastinal Lymph Nodes in PET,
Number analyzed (Participants) | 41
percentage of patients | 44.7 [30.2 to 59.9]

4. Secondary Outcome: Clinical Utility (Avoid More Invasive Procedure)
Description: The clinical utility of puncture under echo-endoscopy puncture has been considered to have a clinical utility, if it allows the patient to avoid more invasive diagnostic procedures (mediastinoscopy or thoracoscopy) or if it allows the patient to benefit from appropriate treatment (result of the malignant biopsy) or to avoid receiving unjustified treatment (result of the benign biopsy): case of patients well classified as malignant/benign by puncture under echo-endoscopy.
  The puncture will be considered to have no clinical utility if the result of the puncture under echo-endoscopy is invalidated by the reference examination, or if the result of the puncture does not allow a diagnosis to be made.
Time Frame: 12 months
Population: Patients evaluable for clinical utility
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Hypermetabolic Mediastinal Lymph Nodes in PET,
Number analyzed (Participants) | 47
percentage of patients | 95.7 [85.46 to 99.48]

5. Other Pre Specified Outcome: Side Effects - Number of Adverse Event Declared According to DINDO Classification
Description: In all cases the side effects associated with the implementation of the guided puncture EUS has been collected and classified according to the classification of surgical complications of Clavien-Dindo [P Clavien and al. Ann Surg 2009, 250: 187-96].
  Classification of surgical complications of Clavien-Dindo ranges from grade 1 (any deviation from the normal postoperative course) to grade 5 (death of patient)
Time Frame: 12 months
Population: Patients with at least one adverse event with Dindo classification (N=38)
Measure: Number; unit: Number of adverse event per grade
Units Other Than Participants: Number of adverse event
Arm/Group | Hypermetabolic Mediastinal Lymph Nodes in PET,
Number analyzed (Participants) | 38
Number analyzed (Number of adverse event) | 68
Number of adverse event per grade
  Not available | 54
  I | 6
  II | 2
  IIIb | 6

ADVERSE EVENTS:
Time Frame: Collection of adverse events (AEs) for 45 days after echo-guided puncture or without time limit if the AE is considered to be related to the puncture, an average of 1 year.
Description: Adverse Event Terms has not been reported in the CRF. AEs related to possible complementary treatments such as chemotherapy has not to been reported in the CRF.
Arm/Group | Hypermetabolic Mediastinal Lymph Nodes in PET,
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 34/47
Other Adverse Events (participants affected / at risk) | 34/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypermetabolic Mediastinal Lymph Nodes in PET, (N=47)
Anemia (Blood and lymphatic system disorders) | 3 (3) — Blood and lymphatic system disorders
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) — Blood and lymphatic system disorders
Heart failure (Cardiac disorders) | 1 (1) — Cardiac disorders
Ascites (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders
General disorders and administration site conditions - Other, specify (General disorders) | 4 (4) — General disorders and administration site conditions
Kidney infection (Infections and infestations) | 1 (1) — Infections and infestations
Urinary tract infection (Infections and infestations) | 1 (1) — Infections and infestations
Fracture (Injury, poisoning and procedural complications) | 1 (1) — Injury, poisoning and procedural complications
Platelet count decreased (Investigations) | 1 (1) — Investigations
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — Metabolism and nutrition disorders
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) — Metabolism and nutrition disorders
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Musculoskeletal and connective tissue disorders
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) — Neoplasms benign, malignant and unspecified (incl cysts and polyps)
Acute kidney injury (Renal and urinary disorders) | 1 (1) — Renal and urinary disorders
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Renal and urinary disorders
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Respiratory, thoracic and mediastinal disorders
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypermetabolic Mediastinal Lymph Nodes in PET, (N=47)
Left inguinal hernia aggravation (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Alteration of the general condition (General disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Ferriprive anemia on melena (Blood and lymphatic system disorders) | 1 (1)
Multifactorial anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Febrile aplasia (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Cervicalgies (Musculoskeletal and connective tissue disorders) | 1 (1)
Surgery for liver metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypoglycemic coma (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Right cruralgia (Nervous system disorders) | 1 (1)
Cryotherapy for pleuropulmonary metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Removal of the left cervical lymph node (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oedemato-ascitic decompensation (Hepatobiliary disorders) | 1 (1) — OEDEMATO-ASCITIC DECOMPENSATION
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Right foot dysesthesia (Nervous system disorders) | 1 (1)
Dysphony (Nervous system disorders) | 1 (1)
Acute dyspney (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysury (Renal and urinary disorders) | 1 (1)
Pulmonary embolisme (Vascular disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile episode (General disorders) | 1 (1)
Extra systole (Cardiac disorders) | 1 (1)
Fracture of the left pubic ramus (Injury, poisoning and procedural complications) | 1 (1)
Hematury (Renal and urinary disorders) | 1 (1)
Hemoptysia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorragia (Vascular disorders) | 4 (4)
Hepatite C (Infections and infestations) | 1 (1)
Hyperkalemy (Metabolism and nutrition disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
Kidney failure (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Laryngospasmus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrale mestastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mucite (Gastrointestinal disorders) | 1 (1)
Mycosis (Infections and infestations) | 1 (1)
Lingual mycosis (Infections and infestations) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Oedeme (General disorders) | 1 (1) — Left lower limb
Oesophagite (Gastrointestinal disorders) | 1 (1)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peritoneal kystic mesotheliome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Disease progression (General disorders) | 1 (1)
Symptomatoc intramedullary progression (General disorders) | 1 (1)
Tumoral progression (General disorders) | 1 (1)
Pyelonephrite with E.COLI and enterobactery (Infections and infestations) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
Lung metastasis resection + lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rhinite (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis of probable urinary origin (Infections and infestations) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)
Cave syndrome and jugular thrombosis (Cardiac disorders) | 1 (1)
Vertebral compression (Musculoskeletal and connective tissue disorders) | 1 (1) — T11 AND L5
Vertebral compression (Musculoskeletal and connective tissue disorders) | 1 (1) — T11, T12 AND L1
Thrombopenia (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Xerophthalmia (Eye disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1)
Aggravation left inguinal hernia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT01892501/Prot_SAP_000.pdf